CLINICAL TRIAL: NCT04208269
Title: A Multilevel Approach to Increasing HPV Vaccine Initiation Among Adolescents - Part 3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB201200143
Record Dates: First submitted 2019-12-19; First posted 2019-12-23 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Human Papilloma Virus
Keywords: preventative; postcard; vaccinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Postcard campaign (Active Comparator)
  Interventions: Other: postcard campaign
- Provider-only intervention (Active Comparator)
  Interventions: Other: Health Information Technology system
- Patient and provider intervention (Active Comparator)
  Interventions: Other: postcard campaign; Other: Health Information Technology system
- Standard care (No Intervention)

INTERVENTIONS:
Other: postcard campaign — Post card sent to parent only
  Arms: Patient and provider intervention; Postcard campaign
Other: Health Information Technology system — Accessed by adolescent and provider only
  Arms: Patient and provider intervention; Provider-only intervention

SUMMARY:
Our project will assess the feasibility and estimate preliminary efficacy of a multilevel intervention to improve HPV vaccine series initiation among adolescents in Medicaid and CHIP. The investigators will use two intervention components: postcards and an iPad survey system. To estimate efficacy the investigators will select potential participants from Florida Medicaid and CHIP. The investigators will assess their claims for the HPV vaccine before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in Florida Medicaid
* Not initiated the HPV vaccine series at the start of the study period.

Exclusion Criteria:

* Anyone who has a severe (life threatening) allergy to any component of HPV vaccine, esp yeast
* Pregnant
* Not enrolled in Florida Medicaid

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 5663 (Actual)
Dates: Start 2013-08-01 (Actual); Primary Completion 2014-04-01 (Actual); Study Completion 2015-03-30 (Actual)

PRIMARY OUTCOMES:
The number of participants receiving HPV vaccine | Up to 5 months
  The percent age eligible participants who initiate HPV vaccination.
Number of preventive care visits | Up to 3 months
  The percent age eligible participants received a preventive care visit

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Staras, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Staras SAS, Vadaparampil ST, Thompson LA, Scherr C, Gurka MJ, Filipp SL, Shenkman EA. Postcard reminders for HPV vaccination mainly primed parents for providers' recommendations. Prev Med Rep. 2020 Aug 26;20:101188. doi: 10.1016/j.pmedr.2020.101188. eCollection 2020 Dec. PMID 32953426